CLINICAL TRIAL: NCT02292641
Title: Investigating the Origins of Pelvic Recurrence in Colorectal Cancer
Brief Title: Beyond TME Origins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Pelican Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCUMAS: 17HH4158
Record Dates: First submitted 2014-05-02; First posted 2014-11-17 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Neoplasms; Adenocarcinoma; Carcinoma
Keywords: Lower Gastrointestinal Tract; Rectum; Diagnostic Imaging; Magnetic Resonance Imaging; Pelvic Exenteration; Neoplasms; Adenocarcinoma; Carcinoma
MeSH Terms: conditions — Neoplasms; Adenocarcinoma; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with pelvic recurrence from primary colorectal cancer (Other): Implementation of imaging assessment proformas describing anatomic pelvic compartments and aetiology of disease recurrence for treatment planning.
  Interventions: Procedure: New Radiological Staging Classification system for patients with advanced and recurrent colorectal cancer undergoing pelvic exenterative surgery

INTERVENTIONS:
Procedure: New Radiological Staging Classification system for patients with advanced and recurrent colorectal cancer undergoing pelvic exenterative surgery — Currently there are no validated criteria or guidelines for judging whether advanced primary or recurrent colorectal cancer can be successfully removed and for selecting which patients should undergo this form of more radical surgery as is exenterative surgery. We are proposing that by validating the detailed evaluation of imaging of the tumour distribution within the pelvis using a new radiological staging classification, this will enable clear selection criteria to be established and will improve surgical planning.

SUMMARY:
All patients with recurrent colorectal cancer in the pelvis are eligible. The original primary tumour staging scans and resected surgical specimen needs to be available. Patients' recurrence will be staged using our proposed MRI classification. We will be assessing the original primary staging scans and histopathology to learn about risk factors for recurrence. We will record treatment for the recurrence, and patients will be followed up for three years.

DETAILED DESCRIPTION:
A prospective and retrospective cohort study to improve surgical and treatment planning using an imaging assessment proforma of advanced and recurrent colorectal cancers. This involves the implementation of imaging assessment proformas describing anatomic pelvic compartments and aetiology of disease recurrence for treatment planning.

ELIGIBILITY:
Inclusion Criteria:

1. Had a primary colorectal adenocarcinoma proven by biopsy taken as part of routine clinical practice
2. Has a confirmed diagnosis of recurrent pelvic colorectal cancer
3. Has previously completed surgical treatment of primary adenocarcinoma of the colon, sigmoid colon or rectum
4. Are able to undergo high resolution MRI for staging prior to treatment decisions
5. Have provided written informed consent to participate in the study
6. Be aged 16 years or over

Exclusion Criteria:

1. Have irresectable extra-pelvic metastatic disease
2. Original baseline staging and preoperative restaging scans (MR for rectal and sigmoid cancers and/or CT for colon and sigmoid cancers) are unavailable
3. Original preoperative, surgical and adjuvant treatment has not been documented or is unavailable

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 383 (Estimated)
Dates: Start 2014-09-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
To change R0 resection rates for locally recurrent rectal cancers with the use of the proposed staging system. | 3 years
  An increase of 20% in R0 resection (from 55% to 75%) for locally recurrent rectal cancers with the use of the proposed staging system

SECONDARY OUTCOMES:
To compare baseline prognostic features against type of recurrence | 3 and 5 years
  Correlation of baseline and post treatment prognostic factors on imaging and pathology against type of recurrence.
To compare the MRI type of recurrence against clinical outcomes | 1, 3 and 5 years
  Proportion of patients with survival >12mths according to type of recurrence as described on MRI
To compare the MRI compartment(s) distribution of recurrence against clinical outcomes | 1, 3 and 5 years
  Proportion of patients with survival >12mths according to compartment(s) of recurrence as described on MRI
To investigate the effect of surgical and non-surgical treatments for recurrence on Quality of Life | 1, 2, 3 and 5 years
  Quality of life assessed using EORTC QLQ-C30
To compare radiology and histopathology compartments in patients undergoing beyond TME surgery for recurrence | Up to 2 years
  The number of compartments predicted as involved on MRI against the number of compartments reported on the corresponding pathology specimens
To measure radiology inter-observer agreement for types of recurrence classification | 5 years
  Kappa agreement between paired radiologists for type of recurrence
To investigate health economic costs of patients with pelvic recurrence against type | Up to 3 years
  Healthcare costs using NHS Reference Costs combined with health resource utilization and QoL data
To map original radiotherapy volumes (including integrated boosts) against types of recurrence | Up to 2 years
  Correlation of dose, type and distribution of radiotherapy against anatomic sites and aetiology of recurrence as seen on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Gina Dr Brown, MD, Principal Investigator — Imperial College London
Locations (4):
- Oslo University Hospital, Oslo, Norway
- United Kingdom (3):
  - St Mark's Hospital, Harrow, London
  - Churchill Hospital, Oxford, Oxfordshire
  - Royal Marsden Hospital NHS Foundation Trust, Sutton